CLINICAL TRIAL: NCT02760394
Title: Hyperbaric Oxygen Therapy in Patients With Chronic Stable Ischemic Heart Disease: An Option for Therapeutic Angiogenesis?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf Harofeh MC (Other Government)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Medical Doctor, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0165-15-ASF
Record Dates: First submitted 2016-04-19; First posted 2016-05-03 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Ischemic Heart Disease
Keywords: chronic ischemic heart disease; coronary bypass; refractory stable angina; HBOT; reperfusion; neoangiogenesis; microvascular; myocardial perfusion
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated group (Active Comparator): 40 daily sessions, 90 minutes of 100% oxygen at pressure of 2 ATA each, five days a week for 8 weeks.
  Interventions: Device: HBOT
- Control group (Other): Following 2 months of follow up the group will be crossed over to receive the same treatment as the treated group
  Interventions: Device: HBOT

INTERVENTIONS:
Device: HBOT — 40 daily sessions, 90 minutes of 100% oxygen at pressure of 2 ATA each, five days a week for 8 weeks.

SUMMARY:
Hyperbaric oxygen therapy (HBOT) is proposed as a possible in vivo angiogenic stimulator for improving microvascular myocardial perfusion and anginal symptoms as assessed by myocardial perfusion imaging and angina questionnaire in patients with chronic stable ischemic heart disease, when no other means to relief symptoms and/or ischemia are available.

DETAILED DESCRIPTION:
Ischemic heart disease is the leading cause of mortality in the United States and second most common in Israel. Myocardial ischemia prevails when imbalance between oxygen demand and delivery to the myocardium occurs: due to increased oxygen demand beyond what can be delivered by increased coronary flow; due to restriction of blood flow from obstruction or stenosis in the coronary circulation in the face of preserved oxygen demand; or combination of these processes. There are two main causes for restricted blood supply to the myocardium: Epicardial atherosclerotic coronary disease or dysfunctional coronary microcirculation. The two processes are often co-occurring in the same patient given the similarities between the risk factors underlying both. As the blood vessels fail to deliver adequate resting or maximal coronary blood flow, either gradually over many years or abruptly during a course of an acute event, myocardial segmental compromise and thus, global cardiac function deteriorates.

The functional hallmark of ischemic left ventricular (LV) segments is their inadequate contractility, manifested as hypokinetic or akinetic segments when examined using either invasive or non-invasive LV functional studies. Ischemic myocardial cells may progress to cellular death, and irreversible scar formation. However, other cells may maintain viability. These viable myocardial segments are of particular clinical importance given their ability to resume contractility with adequate optimal medical therapy and/or revascularization optimization.

Gate SPECT technology allows evaluation of myocardial perfusion and myocardial segmental viability in patients with chronic ischemic heart disease. Studies evaluating the ability of myocardial perfusion studies to predict clinical outcomes are contradictory in that many have shown ability to predict morbidity and mortality endpoints while others didn't .

However, it is intuitively conceivable that invasive and non invasive approaches that are able to reduce ischemic burden as determined by myocardial perfusion imaging, are an important goal for the treatment of patients with chronic ischemic heart disease.

Different standard invasive approaches as percutaneous coronary angioplasty (PCI) and coronary artery bypass grafting (CABG) have been shown to increase myocardial perfusion when serial studies were compared before and after the intervention. Furthermore, non invasive anti-anginal medications as calcium channel blockers, beta blocker and nitrates as well as statins have been shown to similarly produce improvement in myocardial perfusion images as are combinations of these treatments, as required by modern evidence-based guidelines. It is presumed that these non-invasive approaches either decrease myocardial oxygen demand (e.g. Beta blocker) or increase coronary dilation (e.g. Nitrates) as the therapeutic means by which they contribute to ischemia reduction.

During the past decade or so, the concept of "therapeutic angiogenesis" has emerged out of the observation that a significant number of patients are not candidates for standard revascularization procedures or have incomplete revascularization with conventional procedures like PCI or CABG. For example, in patients with two or three vessel coronary artery disease, complete revascularization was successful in 23% and 9% of cases, respectively in one report. The goal of therapeutic angiogenesis is the induction of new coronary arterial vessels that can effectively provide blood supply to the area of myocardium subtended by diseased or occluded native coronary arteries. These "native bypass" vessels could then relieve myocardial ischemia, improve regional and global left ventricular performance, lessen symptoms of angina, and potentially improve patient prognosis. Candidates for pharmacological stimulation of therapeutic angiogenesis in cardiac ischemia include angiogenic cytokines such as Fibroblast Growth Factors (FGF), Vascular Endothelial Growth Factors (VEGF), Hepatocyte Growth /Scatter Factor (HGF/SF), CXC chemokines such as interleukin 8 (IL8) and monocytes chemoattractant protein 1 (MCP-1), growth factors involved in maturation of the vascular tree such as angiopoietins and Platelet Derived Growth Factor (PDGF) and transcription factors that stimulate expression of angiogenic cytokines and their receptors such as Hypoxia-Induced Factor 1α (HIF1α).

Following promising results from pre-clinical and non-controlled studies, several randomized placebo-controlled trials in humans, using some of these candidates, have shown at best, modest clinical endpoints improvement or perfusion enhancing capabilities. Although therapeutic angiogenesis using angiogenesis-enhancing factors is an active research arena, it is still in its infancy and no such strategy have yet achieved acceptance as adjuvant therapy for chronic ischemic heart disease.

In this study, hyperbaric oxygen therapy (HBOT) is proposed as a possible in vivo angiogenic stimulator for improving microvascular myocardial perfusion. Surprisingly, HBOT has not been extensively evaluated in patients with chronic stable ischemic heart disease and to date, its evaluation in cardiovascular diseases was primarily in the context of acute coronary syndrome, amelioration of ischemic-reperfusion injury and stem cell research.

HBOT has been investigated for treatment of numerous diseases for more than 300 years.

The principal effect of HBOT is increasing the solubility of oxygen in plasma to a level sufficient to support tissues with minimal oxygen supply carried on by hemoglobin. Transport of oxygen to mitochondria, the main sites of oxygen utilization within each individual cell, occurs by diffusion, via a stepwise decrease in the driving oxygen pressure gradient. Diffusion oxygen gradient is a vector indicating the direction of the greatest rate of change between oxygen dissolved in the blood and oxygen within the cell/entire tissue. As a whole, breathing oxygen under hyperbaric conditions has been shown to be a potent means of increasing arterial oxygen tension, as well as tissue oxygen tension. For example, at 2 absolute atmospheres (ATA), plasma O2 tension rises above 1110 mmHg, whereas at normal environmental conditions, i.e. at the sea level, it reaches only 98 mmHg. As can be concluded, hyperbaric conditions can provide about a ten-fold increase in the amounts of O2 reaching the hypoxic cardiac tissue. HBO therapy is well tolerated and has been considered safe when used according to the standard protocols, with oxygen pressure not exceeding 3 ATA and treatment sessions limited to a maximum of 120 min.

Multiple studies have suggested that HBOT can enhance angiogenesis but demonstrating enhanced myocardial perfusion (presumably via therapeutic angiogenesis) in humans, have never been attempted. The investigators hypothesized that chronically ischemic viable myocardial tissue is in a state of chronic oxygen demand/delivery imbalance and that physiologic ischemia-induced angiogenesis during regenerative/repair processes, aimed to restore oxygen delivery, has been "burned out". Since all the regenerative/repair processes have common denominator: they are all energy/oxygen dependent, it might be possible that HBOT can enables the metabolic changes needed to reignite those regeneration processes, simply by supplying the missing energy/oxygen.

Method:

After signing the informed consent, patients will be randomized in 1:1 manner into the treated or the control-cross group. After the randomization, patients will be invited for baseline evaluation that included full review of their medical status and complete physical examination. Patients will be instructed to refrain from any changes in their chronic medications or life style (e.g. exercise regimen) and to avoid new medications unless clinically indicated and approved by the study investigators. Quality of life (QOL) assessments (Seattle Angina Questionnaire [SAQ] translated to Hebrew) will be completed at baseline and every 2 month in the control period or following the treatment period.

After their inclusion, all patients will undergo baseline myocardial perfusion study. Afterwards, patients will be randomized to two groups: a treated group and a cross group. Patients in the treated group will undergo HBOT treatment for 2 months and after that will repeat the same-protocol myocardial perfusion study and questionnaire, before entering a 2 month control period. Patients in the cross group will be evaluated at baseline, after a 2 month control period of no treatment and after 2 month period of HBOT treatment (after the cross to HBOT).

The following HBOT treatment protocol will be practiced: 40 daily sessions, 90 minutes of 100% oxygen at pressure of 2 ATA each, five days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older.
* Symptomatic or asymptomatic chronic ischemic heart disease patients, with no more than moderate systolic dysfunction (EF>30%) on optimal medical treatment who have been evaluated for myocardial ischemia using myocardial perfusion study and coronary angiography.
* Patients who demonstrate significant myocardial perfusion defect, defined as ≥5% global perfusion defect and/or ≥3 segments with perfusion defect out of 17 myocardial segments, and were found to have coronary artery disease not amenable for PCI or CABG (or re-CABG) due to anatomical or medical considerations.
* Clinical stable patients in the 3 months before randomization. Good functional class as determinate by the New York Heart association functional status I-III and Canadian Cardiovascular Society Angina class I-III. Optimal medical therapy defined by chronic regular use of a combination of more than 3 antianginal medications (beta blockers, calcium channel blockers, nitrates, unless contraindicated for any reason) and/or secondary prevention drugs (aspirin, aldosterone antagonists, angiotensin converting enzyme inhibitors, angiotensin receptor blockers, statins, unless contraindicated for any reason).

Exclusion Criteria:

* Current smokers or smoking patients who could not comply with the demand to cease smoking prior to inclusion.
* Had been treated with HBOT for any other reasons prior to their inclusion
* Have any other indication for HBOT;
* Chest pathology incompatible with pressure changes;
* Inner ear disease;
* Patients suffering from claustrophobia;
* Inability to sign written informed consent.
* Patients unable to perform exercise tolerance test for any reason
* Hospital admission due to acute coronary syndrome or congestive heart failure exacerbation in the past 3 month before randomization
* r CCS class IV angina
* Patients currently in NYHA functional class IV
* Severe or uncontrolled other medical illness as advanced liver, kidney or oncologic diseases

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
change in percentile fixed and reversible defects in myocardial perfusion imaging results | 2 months
  The myocardial perfusion images will be analyzed at baseline and at the end of treatment and control periods to include both percentile of fixed defects and percentile of reversible defects. The images will undergo computerized processing in order for the pre-post images to be comparable.

SECONDARY OUTCOMES:
change in symptoms using the Seattle Angina Questionnaire | 2 months
  Symptoms will be evaluated using the Seattle Angina Questionnaire during baseline and following control and treatment periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No